CLINICAL TRIAL: NCT04794894
Title: Wellness and Quality of Life Perceptions of People With Traumatic Brain Injury Receiving Post-acute Telerehabilitation Versus Clinic-based Services
Brief Title: Wellness and Quality of Life Perceptions of People With Traumatic Brain Injury
Status: Enrolling by invitation | Type: Observational
Sponsor: Quality Living, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: Tele Wellness
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Brain Injuries, Traumatic
Keywords: Therapy; Health-related Quality of Life
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telerehabilitation services: Physical therapy, occupational therapy, speech-language therapy, and/or counseling provided at home via telecommunication technologies.
  Interventions: Behavioral: outpatient rehabilitation
- Clinic-based rehabilitation services: Physical therapy, occupational therapy, speech-language therapy, and/or counseling provided at a local facility.
  Interventions: Behavioral: outpatient rehabilitation

INTERVENTIONS:
Behavioral: outpatient rehabilitation — Treatment provided after completion of inpatient, acute rehabilitation.

SUMMARY:
Telerehabilitation is a service delivery method that has grown substantially in recent years. It has both advantages and disadvantages in comparison to clinic-based services. For example, telerehabilitation is advantageous for people residing in locations in which specialized rehabilitation services are scarce; however, it has the disadvantage of being dependent on reliable internet connections that are not available in all locations. Also, some people prefer the privacy afforded by receiving treatment in their home, but other people prefer the interaction with other clients with similar challenges afforded by attending sessions in clinic-based settings. Other questions about advantages and disadvantages of telerehabilitation remain unexplored. One such question is the focus of this research and concerns the effect of receiving post-acute telerehabilitation services versus clinic-based services on the general well-being and quality of life experienced by people with traumatic brain injury. The study purpose is to compare changes in wellness and quality of life occurring over a four-month period during which people with traumatic brain injury receive post-acute services either via telerehabilitation or at an outpatient facility.

ELIGIBILITY:
Inclusion Criteria:

* Sustained traumatic brain injury
* Receiving inpatient services at Quality Living, Inc., Omaha, NE
* Fluent in English
* Scheduled to receive either telerehabilitation or clinic-based rehabilitation services after discharge from Quality Living, Inc.

Exclusion Criteria:

* Receiving services on a scholarship basis from Quality Living, Inc., Omaha, NE
* Scheduled to receive a combination of telerehabilitation and clinic-based services after discharge from Quality Living, Inc.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty adults with traumatic brain injury will comprise the participant sample. Prospective participants will be from a convenience sample of people with traumatic brain injury nearing discharge from Quality Living's inpatient program. Participants will form two subgroups-those whose prospective outpatient treatment will be through clinic-based services from practitioners near their home and those whose continued rehabilitation will be through telerehabilitation services. Each person's decision about clinic-based versus telerehabilitation service will stem from factors including funding, local availability and access, individual preference, and treatment team recommendations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Quality of Life after Brain Injury | Change from baseline at 4 months
  37-item questionnaire designed to measure six health-related quality of life dimensions for people with TBI
Changes in Outlook - Short | Change from baseline at 4 months
  10-item self-report instrument assessing both positive and negative reactions to adversity and traumatic experiences.
Generalized Anxiety Disorder Screener - 7 | Change from baseline at 4 months
  7-item self-report instrument designed to screen for symptoms and severity of generalized anxiety in adults.
Beck Depression Inventory - II | Change from baseline at 4 months
  21-item self-report instrument on which people rate their experience with depression symptoms within the past two weeks.

SECONDARY OUTCOMES:
Telerehabilitation or Clinic-based Post-acute Treatment Survey | 4 months after study enrollment
  Researcher-designed survey to capture perceptions about treatments received. It includes 2 questions about the length and intensity of physical therapy, occupational therapy, speech-language therapy, and counseling/psychology services and 15 items about the convenience, focus, and outcome of treatment as well as the quality of the therapist-client relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hux, Ph.D., Principal Investigator — Quality Living, Inc.
Locations (1):
- Quality Living, Inc., Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No